CLINICAL TRIAL: NCT06621576
Title: First-in-Human Pilot Study of Epicardial Circular RNA-HM2002 Injection in CABG for Ischemic Heart Failure
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai CirCode Biomed Co.,Ltd (Industry); Shanghai Bestudy Medical Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and Director, Department of Cardiac Surgery, Vice President, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM2002-001
Record Dates: First submitted 2024-09-17; First posted 2024-10-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Ischaemic Heart Disease; Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HM2002 Injection group (Experimental): First sentinel enrollment, no DLT events followed by re-enrollment after 2 cases
  Interventions: Drug: HM2002 injection

INTERVENTIONS:
Drug: HM2002 injection — Eligible subjects under general anesthesia will undergo CABG surgery. After completing the distal anastomosis, 5mg of HM2002 injection solution drawn into a 1 ml syringe will be administered via multi-point injection using an OT needle or insulin needle (preferably a 30G needle). The injections will be spaced approximately 1 cm apart, with no more than 30 injection points, into the myocardium at the edge of the MI area (with obvious infarcts) or the area of the diseased coronary artery branches (without obvious infarcts) through the epicardium.

SUMMARY:
This exploratory, single-center, open-label clinical trial assesses the safety, tolerability, and potential efficacy of a single 5 mg dose of HM2002 injection administered via multiple-point epicardial injections for treating ischemic heart failure. Three patients aged 18-80 undergoing elective coronary artery bypass grafting (CABG) surgery will participate. Using a sentinel dosing approach, the first subject will receive HM2002, followed by a 14-day safety observation before dosing the remaining participants. If any serious adverse events or dose-limiting toxicities occur in the first subject, a Safety Review Committee will evaluate the safety data to determine whether to continue or terminate the trial.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-dose, open-label investigator-initiated exploratory clinical trial (IIT study) designed to evaluate the safety, tolerability, and potential clinical efficacy of the exploratory dose HM2002 injection administered via single-dose, multiple-point injections through the epicardium for the treatment of ischemic heart failure. The study plans to enroll three patients aged between 18 and 80 years who are scheduled to undergo elective coronary artery bypass grafting (CABG) surgery and have ischemic heart failure. Eligible patients will become study subjects after providing full written informed consent and successfully passing the inclusion and exclusion criteria screening. The exploratory dose for this trial is 5 mg HM2002 injection. The three subjects will be dosed following the sentinel dosing principle. Specifically, after the first subject completes dosing, there will be a minimum interval of 14 days (2 weeks) to confirm safety and tolerability before enrolling the remaining two subjects. If any serious adverse event (SAE) or dose-limiting toxicity (DLT) occurs in the first subject, a Safety Review Committee (SRC) meeting will be convened to review all collected safety data. The committee will then determine whether to proceed with the enrollment of subsequent subjects or terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria:

1. be ≥18 and ≤80 years of age at the time of signing the informative and be of either sex;
2. have ischemic heart failure (IHF) with left ventricular ejection fraction (LVEF) ≤50% by echocardiography (ECHO), New York Heart Association (NYHA) cardiac function class 3-4, and be proposed to undergo elective coronary artery bypass grafting (CABG);
3. voluntarily sign the informed consent form and fully understand the content, process and possible adverse reactions of the trial. Be able to complete the study according to the requirements of the trial protocol and have good compliance;

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from this study:

1. subjects with the following concomitant symptoms or diseases:

   1. ECHO-confirmed LVEF ≤ 20%;
   2. History of malignant arrhythmias (including multiple ventricular pre-systole, premature ventricular dystocia, tricyclic rhythm, or ventricular tachycardia) manifesting symptomatically or requiring treatment (CTCAE grade 3);
   3. atrial fibrillation (including paroxysmal atrial fibrillation);
   4. Long QT syndrome;
   5. Estimated glomerular filtration rate (eGFR) ≤ 30 mL/min/1.73 m2; f. Serum gammaglutamyl (GGT) ≤ 1.5 mL/min/1.73 m2
   6. Serum alanine aminotransferase (ALT) or aminotransferase (AST) > 3 x upper limit normal (ULN) and total bilirubin (TBIL) > 2 x ULN or more;
   7. Severe coagulation disorders, bleeding disorders, etc;
   8. history of active human immunodeficiency virus (HIV), active hepatitis C virus (HCV), or active hepatitis B virus (HBV); active HIV, HCV, and HBV infections are defined as:

   <!-- -->

   1. HIV antibody positive;
   2. Anti-HCV antibody and positive for HCV RNA;
   3. HBsAg positive and HBV DNA ≥1000 cps/ml (or 200 IU/ml); i. current malignancy, or a history of malignancy.
2. need for concurrent cardiac or non-cardiac interventional or surgical procedures other than CABG (e.g., valve surgery, ventricular wall tumor surgery, peripheral arterial stenting or surgery)
3. patients with prior systemic or cardiac therapy with similar nucleic acid medications
4. a known history of drug abuse or drug allergy
5. pregnant or lactating women or those who are not using effective contraception;
6. other circumstances judged by the investigator to be inappropriate, such as the investigator's judgment that the subject may be exposed to substantial safety risks, or interference with the results of the study, or lack of participation in completing this trial in accordance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs) and Clinically Meaningful Changes from Baseline in Clinical Laboratory Tests, Vital Signs, and Electrocardiogram Parameters | 6 months
  To assess the safety of a single 5 mg dose of HM2002 injection in treating ischemic heart failure by evaluating the incidence of adverse events (AEs) and serious adverse events (SAEs) as categorized according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, along with clinically meaningful changes from baseline in clinical laboratory tests (including complete blood count [CBC], liver function tests [LFTs], renal function tests [RFTs], and coagulation function), vital signs (such as systolic and diastolic blood pressure, heart rate, respiratory rate, and body temperature), and 12-lead electrocardiogram (ECG) parameters (including heart rhythm disturbances, ST segment deviations, T wave abnormalities, and alterations in PR or QT interval).

SECONDARY OUTCOMES:
Myocardial Perfusion Changes | Baseline, 6 months
  Changes in blood perfusion of the ischemic myocardial injection segments measured by resting cardiac magnetic resonance (CMR) perfusion imaging
CMR Assessment of LVEF | Baseline, 6 months
  Changes in LVEF assessed by CMR
NT-proBNP Level Changes | Baseline, 1 month, 3 months, and 6 months
  Changes in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels
Echocardiographic Assessment of Cardiac Function | Baseline, 1 month, 3 months, and 6 months
  Changes in Left Ventricular Ejection Fraction (LVEF) assessed by echocardiography
Perfusion Changes in Ischemic Myocardium | Baseline, 6 months
  Changes in perfusion of the ischemic myocardial injection segments measured by SPECT
Metabolism Changes in Ischemic Myocardium | Baseline, 6 months
  Changes in metabolism of the ischemic myocardial injection segments measured by PET
Angina Score Changes | Baseline, 1 month, 3 months, and 6 months
  Changes in angina score measured by the Seattle Angina Questionnaire (SAQ), ranging from 0 to 100 per domain, with higher scores indicating a better outcome.
Quality of Life Changes | Baseline, 1 month, 3 months, and 6 months
  Changes in quality of life (QoL) assessed by the Minnesota Living with Heart Failure Questionnaire (MLHFQ), ranging from 0 to 105, with higher scores indicating a worse outcome.
NYHA Functional Classification Changes | Baseline, 1 month, 3 months, and 6 months
  Changes in New York Heart Association (NYHA) functional classification. The NYHA classification ranges from Class 1 to 4. Higher scores (Class 4) indicate worse functional status, while lower scores (Class 1) indicate better functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Principal Investigator — Ruijin Hospital; Yunpeng Zhu, MD, Study Director — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China